CLINICAL TRIAL: NCT03954483
Title: Measurement of the Hippocampal Theta Rhythm From the Outer Ear Canal
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Zeinab Dastgheib, Principal Investigator, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: B2018:096
Record Dates: First submitted 2019-05-14; First posted 2019-05-17 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Buspirone; Tablets; Triazolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Buspirone (Experimental): Participants will receive buspirone 10 mg prior to experiments.
  Interventions: Drug: Buspirone 10 Mg Oral Tablet
- Triazolam (Experimental): Participants will receive triazolam 0.25 mg prior to experiments.
  Interventions: Drug: Triazolam 0.25 MG Oral Tablet
- Placebo (Placebo Comparator): Participants will receive a placebo prior to experiments.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Buspirone 10 Mg Oral Tablet — Orally administered prior to experiments.
  Arms: Buspirone
Drug: Triazolam 0.25 MG Oral Tablet — Orally administered prior to experiments.
  Arms: Triazolam
Drug: Placebo oral tablet — Orally administered prior to experiments.
  Arms: Placebo

SUMMARY:
New technologies are needed to help diagnose anxiety disorders. EVestG has facilitated the identification of numerous possible biomarkers of several psychiatric disorders. Some EVestG features seem to be caused by differences in low-frequency modulation that is consistent (both in frequency and behaviour) with the hippocampal rhythm (theta), which is known to play a role in anxiety. Critically, there is ample support in the literature for an anatomical and functional basis for the modulation of vestibular signals via theta. If anxiety could be measured continuously, perhaps throughout a patient's day, or throughout a task, it might be able to confirm an anxiety disorder. However, current techniques for measuring theta are highly invasive, performed rarely, and only in epilepsy patients. EVestG technology, however, is non-invasive, and could potentially record anxiety levels in any subject for extended periods of time. The proposed study will attempt to identify hippocampal theta in vestibular signals in healthy participants through a double-blind administration of two different drugs that are dissimilar both pharmacologically and in acute clinical effects but which are known to reduce the theta rhythm.

DETAILED DESCRIPTION:
OBJECTIVE:

To investigate whether the gross electrical activity of the outer ear canal contains the hippocampal theta rhythm (theta) - a potential biomarker for anxiety - and to identify potential modulatory effects that theta may have on vestibular signals, using electrovestibulography (EVestG).

STUDY POPULATION:

Forty-two (42) individuals, aged between 18 and 40 years, who report no psychological treatment in the past year.

The means of recruiting participants will conform with University of Manitoba Research Ethics Board guidelines. All participants will provide written, informed consent prior to participation. Additional consent for the drug experiment will be provided by a physician on the research team who will also write prescriptions for the study drugs.

STUDY DESIGN:

Forty-two (42) participants will be randomly allocated to one of three parallel groups (of equal size): The 'triazolam group,' in which participants will receive 0.25 mg of (oral) triazolam prior to the experiments; the 'buspirone group,' in which participants will receive 10 mg of (oral) buspirone prior to the experiments; and the 'placebo group,' in which participants will receive a placebo pill prior to the experiments.

The study will consist of two experiments: "Whole-Body Motion" (WBM); and the "Stop Signal Task" (SST). Throughout these experiments, Electroencephalography (EEG) activity will be simultaneously recorded from the outer ear canal, (via EVestG electrodes), and the frontal F7, Fz and F8 sites, (using a minimalist configuration of surface electrodes).

All participants who meet inclusion criteria and provide informed consent will participate in these experiments and complete a series of tests at the Riverview Health Centre, over a period of approximately 2-3 hours. These tests include: an audiogram and a balance test; as well as a series of questionnaires that screen for depression and assess cognition, symptom severity, fatigue and balance. The procedure may also include frontal brain asymmetry measures via surface electrode EEG recordings.

HYPOTHESES:

In the SST experiment, the WBM experiment, and resting states (between rotations), we hypothesize that for the three study groups: 1) any 4-12 Hz modulation of vestibular field potentials will be lowest (in frequency) in the drug groups and highest in the placebo group; 2) the drug groups will have EEG spectral peaks in the 4-12 Hz range that are the lowest (in frequency) while the placebo group peaks will be the highest; 3) overall 4-12 Hz EEG power will be lowest in the drug groups and highest in the placebo group; 4) in general, 4-12 Hz EEG activity and 4-12 Hz entrainment of EVestG field potentials (FPs) will be most prominent and occur most often in the placebo group and least often in the drug groups.

The placebo group is expected to show the highest degree of theta-range coherence between mPFC and outer ear canal activity, especially during WBM movements and intermediate delay SST Stop trials, but also during resting state. The drug groups are predicted to exhibit the lowest degree of this coherence.

Theta frequency is expected to correlate with state anxiety to the degree that it will separate high- and low-scoring individuals on the State-Trait Anxiety Inventory (STAI) test. It is hypothesized that trait anxiety, (also measured by the STAI test), will correlate with features unrelated to theta but similar to those identified in previous EVestG studies that involved depressed patients, where differentiating features were found in average FP waveforms.

METHODOLOGY:

Note: During the COVID-19 pandemic, some of the procedures in this section will be modified. (Please see Appendix A of the protocol for standard operating procedures during the Covid-19 pandemic).

Participants will have the details of the study explained to them before they sign a written consent form. They will then be given the (2-minute) Standing Balance Test (SBT) and the (5-minute) Audiogram. [Any subjects that fail the SBT will be given the (5-minute) Vestibular Disorders Activities of Daily Living Scale (VADL) questionnaire, and subjects who fail the VADL or Audiogram will be excluded]. They will then receive a capsule that contains either 0.25 mg of triazolam, 10 mg of buspirone, or a placebo pill, where the contents of the capsule will be randomly determined by a computer code. Next, they will complete a series of tests and questionnaires. First, the (5-minute) Barnes Akathisia Rating Scale (BARS) and (1-minute) Stanford Sleepiness Scale (SSS) will be conducted. Next, they will complete the (10-minute) Montreal Cognitive Assessment (MOCA) test before filling out both the (10-minute) Eysenck Personality Questionnaire - Revised (EPQ-R) and (10-minute) Spielberger State-Trait Anxiety Inventory (STAI) questionnaires. Some of the questionnaires will be administered by a computer program.

Prior to the experiments, head circumferences will be measured, and electrodes will be attached at F7, Fz and F8 (for analysis) and AFz (Electro Cap Int. Gnd), according to the international 10/20 system; as well as above, below, and to the right of the right eye, and to the left of the left eye; and on both mastoids; with impedances lowered to below 5 kΩ. Next, EVestG electrodes will be positioned, (as per Section 4.3 of the protocol). Electrocardiogram electrodes may also be employed near the wrists/ankles. Participants will then be led to the hydraulic chair that they will remain seated in during the experiments. The abovementioned tests, questionnaires and electrode placements should take about 1 hour.

The first experiment is the SST (see Section 4.15 of the protocol), for which the hydraulic chair will remain motionless. A laptop will be placed in front of the participant. The SST takes roughly 15 minutes to complete.

The second experiment consists of whole-body rotations and translations in the hydraulic chair, (as described in Section 4.3). Each movement will be performed twice, with four different motions from the sitting upright position and two from the supine position. This experiment should take about 30 minutes.

Next, the STAI questionnaire will be administered again, and participants will be screened for depression and cognitive decline with the (15-minute) Montgomery Asberg Depression Rating Scale (MADRS) and (10-minute) Mini-Mental State Examination (MMSE), respectively. The (15-minute) Mini-Internal Neuropsychiatric Interview (M.I.N.I.) will also be used to screen for symptoms.

Finally, all electrodes, tape and superficial gel will be removed from the participant, whom the investigator will encourage to wash their ears with warm water as soon as possible. A total of 2-3 hours will have passed since the capsule was taken. Participants will remain on the fourth floor of the Administration Building at RHC and will be monitored until any drug effects will have worn off. They will be reminded not to operate a motor vehicle to return home and will have arranged an alternate mode of transportation beforehand and will be provided a data sheet for the drug they received.

STATISTICAL ANALYSIS:

Statistical analyses will include MANOVAs and t-tests on power spectra from EVestG and EEG recordings to look for differences between groups. Correlation measures will be used to identify coherence between EVestG and EEG recordings, as well as between symptom rating scores and spectra from EVestG and EEG recordings.

ELIGIBILITY:
Inclusion Criteria:

• Males and females who are between 18 and 40 years of age.

Exclusion Criteria:

* Psychological treatment in the past year or taking any psychiatric drug.
* Drugs that interact with the study drugs or that have anxiolytic/anxiogenic properties.
* Antibiotics or natural health products that inhibit/induce CYP3A4 or CYP2D6.
* History of substance use disorder or family history of substance use disorder.
* Pregnancy (or breastfeeding), left handedness, or colour blindness.
* Individuals who have a current diagnosis, or history of, a neurological illness.
* A history of stroke, head injury, loss of consciousness, epilepsy.
* Kidney or liver disease/impairment.
* COPD or sleep apnea.
* Skin lesions involving the ear canal, self-reported or as assessed in examination at the lab.
* Any unknown balance disorders, as assessed by investigator via balance test.
* Major hearing loss, self-reported or as assessed by investigator via audiogram.
* Allergic skin reactions to chemical agents including detergents.
* Heart disease, lung disease or diabetes.
* Influenza, Covid-19, or flu-like symptoms.
* Recovering from an accident, injury, or operation.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
EEG power spectrum | Derived from EEGs recorded for 30-45 mins
  4-12 Hz EEG power spectrum at F8 (10/20 international system) and in outer ear canal.
4-12 Hz modulation | Derived from EEGs recorded for 30-45 mins.
  4-12 Hz modulation of field potentials recorded in outer ear canal.

SECONDARY OUTCOMES:
Signal correlations | Derived from EEGs recorded for 30-45 mins
  4-12 Hz correlations between F8 (10/20 international system) and outer ear canal activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Riverview Health Centre, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No
Data might be shared in the future.